CLINICAL TRIAL: NCT05873920
Title: Impact of Individual Atrial Arrhythmia Substrate on the Outcome Following Radiofrequency-Guided Catheter Ablation for Atrial Fibrillation in Patients With Diabetes Mellitus
Brief Title: Atrial Fibrillation and Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heart and Diabetes Center North-Rhine Westfalia (Other)
Responsible Party: Sponsor
Other Study IDs: HDZ-ER_004_DG
Record Dates: First submitted 2023-05-16; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Atrial Fibrillation; Arrhythmias, Cardiac; Heart Diseases; Cardiovascular Diseases; Pathologic Processes
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Heart Diseases; Cardiovascular Diseases; Pathologic Processes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Single center prospective study to analyze the impact of diabetes mellitus on patients' outcome following radiofrequency-guided catheter ablation for atrial fibrillation.

DETAILED DESCRIPTION:
A total number of 50 patients with diabetes mellitus will undergo radiofrequency-guided catheter ablation for atrial fibrillation. Pre-procedural cardiac MRI will be performed with late-gadolinium enhancement to visualize the individual amount and distribution of fibrosis in the right and left atrium. The relationship between diabetes mellitus and individual atrial arrhythmia substrates as well as patients' outcome following catheter ablation will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing their 1st radiofrequency-guided catheter ablation for atrial fibrillation
* Diabetes mellitus
* Able to understand and willing to sign the Informed Consent Form.
* Age ≥18 years.

Exclusion Criteria:

* Contraindication for DE-MRI with a full dose of gadolinium-based contrast agent.
* Previous left atrial ablation or surgical procedure
* Women currently pregnant, breastfeeding, or of childbearing age not currently taking or not willing to use a reliable form of contraception
* Mental or physical inability to take part in the study
* Morbid obesity (BMI > 35), or inability to be placed in MRI due to body mass.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 50 consecutive patients with diabetes mellitus and symptomatic atrial fibrillation will be included in this prospective observational analysis. All patients will be treated for atrial fibrillation at the Heart and Diabetes Center NRW, Bad Oeynhausen, Germany. Written informed will be obtained from each patient, the study concept complies with the Declaration of Helsinki and the institutional review board already approved the study design. Catheter ablation will be performed under deep sedation. In all patients preprocedural magnetic resonance imaging (MRI) will be performed prior to the intervention to visualize the individual amount and distribution of fibrosis and to visualize the anatomical location and course of the esophagus.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
atrial fibrillation recurrence | 12 months
  atrial fibrillation recurrence following catheter ablation

CONTACTS AND LOCATIONS:
Locations (1):
- Herz- und Diabeteszentrum NRW, Bad Oeynhausen, Germany